CLINICAL TRIAL: NCT04376203
Title: What is the Relation of Microbiome to Papillary Thyroid Microcarcinoma Development?
Brief Title: Microbiome and Papillary Thyroid Microcarcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Stefanos Stefanou, MD, University of Ioannina
Other Study IDs: Endocrine surgery Unit UOI 1
Record Dates: First submitted 2020-05-02; First posted 2020-05-06 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Papillary Thyroid Microcarcinoma; Microbiome
Keywords: Microbiome; Papillary Thyroid Microcarcinoma
MeSH Terms: conditions — Papillary Thyroid Microcarcinoma | interventions — Thyroidectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: any patient with indications for thyroidectomy other than confirmed preoperative cancer
  Interventions: Procedure: Thyroidectomy
- Thyroid microcarcinoma: either preoperative detection or random finding after thyroidectomy of another indication.
  Interventions: Procedure: Thyroidectomy

INTERVENTIONS:
Procedure: Thyroidectomy — Typical Thyroidectomy

SUMMARY:
It has been shown that gut microbiome and microbiome metabolism can regulate or control the initiation of a cancer process. To the best of the investigators knowledge, no study has directly shown the relationship of the thyroid microcarcinoma to the human microbiome. In this work, the aim is to detect the microbiome in peripheral blood in a patient with a thyroid gland carcinoma, and to correlate it with the disease, compared to the microbiome of a group of patients who did not find another thyroid gland carcinoma

DETAILED DESCRIPTION:
Measurements of biological markers and tumor cell motility may be useful in predicting early whether a papillary thyroid microcarcinoma (PTMC) will develop to invasive carcinoma. Ideally, patients at high risk of progression may undergo immediate surgery instead of active surveillance and those with a very low likelihood of tumor progression may be included in an active surveillance protocol. Future research should focus on the development of new predictive early markers of papillary thyroid carcinoma during patient follow-up. From the above, it is clear the need to develop a new marker that raises the suspicion of possible thyroid microcarcinoma, if it is not preoperatively detected by the needle biopsy method and the patient has the indication for surgery for another benign thyroid disease. To date, there are no absolute biological and clinical parameters distinguishing a low risk from a high risk PTMC. If the fine needle aspiration shows stage V and VI Bethesda classification, and there is a high suspicion of PTMC, then questions such as the extent of the surgery, lobectomy or total thyroidectomy are beginning to be raised. The next dilemma is lymphadenectomy. The dilemma is greater if there are enlarged cervical lymph nodes (diameter over 1 cm in diameter of the small axis) and subsequently micromestases are confirmed. Another entity is when the cervical lymph nodes are not pathologically enlarged. This clinical situation is often emphasized as 60-80% of PTMC patients have metastases. By correlating a possible difference in the microbiome of a participants peripheral blood preoperatively, together with the imaging data, there may have been another marker of early PTMC detection and patient management planning respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are going to have surgery for some thyroid disease, benign or malignant

Exclusion Criteria:

* Recent, less than 3 months, infection of any system
* Receiving antibiotic or antiviral medication in the previous trimester
* Patient with chronic virus or bacterial infection
* Patient with dermatological disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients with indication for surgery for thyroid disease
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-07-27 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Type of microbiome in peripheral blood sample of a patient with papillary thyroid microcarcinoma | preoperatively periferal blood collection, perioperatively periferal blood colection
  Microbiome in a sample of peripheral blood in a patient with PTMC and to correlate it with the disease as a diagnostic marker compared to patients without any type of thyroid cancer.

CONTACTS AND LOCATIONS:
Overall Officials: KONSTANTINOS VLACHOS, Associate Professor of Surgery, Study Chair — University of Ioannina; IOANNIS KOUTELIDAKIS, Associate Professor of Surgery, Study Chair — Aristotle University Of Thessaloniki

IPD SHARING:
Plan to Share IPD: Yes
all data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Available in one year and for 3 years long

REFERENCES:
- [Background] Caporaso JG, Lauber CL, Costello EK, Berg-Lyons D, Gonzalez A, Stombaugh J, Knights D, Gajer P, Ravel J, Fierer N, Gordon JI, Knight R. Moving pictures of the human microbiome. Genome Biol. 2011;12(5):R50. doi: 10.1186/gb-2011-12-5-r50. PMID 21624126
- [Background] Choi JB, Lee WK, Lee SG, Ryu H, Lee CR, Kang SW, Jeong JJ, Nam KH, Lee EJ, Chung WY, Jo YS, Lee J. Long-term oncologic outcomes of papillary thyroid microcarcinoma according to the presence of clinically apparent lymph node metastasis: a large retrospective analysis of 5,348 patients. Cancer Manag Res. 2018 Aug 27;10:2883-2891. doi: 10.2147/CMAR.S173853. eCollection 2018. PMID 30214283
- [Background] David LA, Maurice CF, Carmody RN, Gootenberg DB, Button JE, Wolfe BE, Ling AV, Devlin AS, Varma Y, Fischbach MA, Biddinger SB, Dutton RJ, Turnbaugh PJ. Diet rapidly and reproducibly alters the human gut microbiome. Nature. 2014 Jan 23;505(7484):559-63. doi: 10.1038/nature12820. Epub 2013 Dec 11. PMID 24336217
- [Background] Feng J, Zhao F, Sun J, Lin B, Zhao L, Liu Y, Jin Y, Li S, Li A, Wei Y. Alterations in the gut microbiota and metabolite profiles of thyroid carcinoma patients. Int J Cancer. 2019 Jun 1;144(11):2728-2745. doi: 10.1002/ijc.32007. Epub 2018 Dec 24. PMID 30565661
- [Background] Frank DN, St Amand AL, Feldman RA, Boedeker EC, Harpaz N, Pace NR. Molecular-phylogenetic characterization of microbial community imbalances in human inflammatory bowel diseases. Proc Natl Acad Sci U S A. 2007 Aug 21;104(34):13780-5. doi: 10.1073/pnas.0706625104. Epub 2007 Aug 15. PMID 17699621
- [Background] Gevers D, Kugathasan S, Denson LA, Vazquez-Baeza Y, Van Treuren W, Ren B, Schwager E, Knights D, Song SJ, Yassour M, Morgan XC, Kostic AD, Luo C, Gonzalez A, McDonald D, Haberman Y, Walters T, Baker S, Rosh J, Stephens M, Heyman M, Markowitz J, Baldassano R, Griffiths A, Sylvester F, Mack D, Kim S, Crandall W, Hyams J, Huttenhower C, Knight R, Xavier RJ. The treatment-naive microbiome in new-onset Crohn's disease. Cell Host Microbe. 2014 Mar 12;15(3):382-392. doi: 10.1016/j.chom.2014.02.005. PMID 24629344
- [Background] Grice EA, Segre JA. The skin microbiome. Nat Rev Microbiol. 2011 Apr;9(4):244-53. doi: 10.1038/nrmicro2537. PMID 21407241
- [Background] Grice EA, Kong HH, Conlan S, Deming CB, Davis J, Young AC; NISC Comparative Sequencing Program; Bouffard GG, Blakesley RW, Murray PR, Green ED, Turner ML, Segre JA. Topographical and temporal diversity of the human skin microbiome. Science. 2009 May 29;324(5931):1190-2. doi: 10.1126/science.1171700. PMID 19478181
- [Background] Hannigan GD, Meisel JS, Tyldsley AS, Zheng Q, Hodkinson BP, SanMiguel AJ, Minot S, Bushman FD, Grice EA. The human skin double-stranded DNA virome: topographical and temporal diversity, genetic enrichment, and dynamic associations with the host microbiome. mBio. 2015 Oct 20;6(5):e01578-15. doi: 10.1128/mBio.01578-15. PMID 26489866
- [Background] Hedinger C, Williams ED, Sobin LH. The WHO histological classification of thyroid tumors: a commentary on the second edition. Cancer. 1989 Mar 1;63(5):908-11. doi: 10.1002/1097-0142(19890301)63:53.0.co;2-i. PMID 2914297
- [Background] Ishaq HM, Mohammad IS, Shahzad M, Ma C, Raza MA, Wu X, Guo H, Shi P, Xu J. Molecular Alteration Analysis of Human Gut Microbial Composition in Graves' disease Patients. Int J Biol Sci. 2018 Sep 7;14(11):1558-1570. doi: 10.7150/ijbs.24151. eCollection 2018. PMID 30263008
- [Background] Kaliszewski K, Diakowska D, Wojtczak B, Forkasiewicz Z, Pupka D, Nowak L, Rudnicki J. Which papillary thyroid microcarcinoma should be treated as "true cancer" and which as "precancer"? World J Surg Oncol. 2019 May 31;17(1):91. doi: 10.1186/s12957-019-1638-0. PMID 31146753
- [Background] Kasaikina MV, Kravtsova MA, Lee BC, Seravalli J, Peterson DA, Walter J, Legge R, Benson AK, Hatfield DL, Gladyshev VN. Dietary selenium affects host selenoproteome expression by influencing the gut microbiota. FASEB J. 2011 Jul;25(7):2492-9. doi: 10.1096/fj.11-181990. Epub 2011 Apr 14. PMID 21493887
- [Background] Koenig JE, Spor A, Scalfone N, Fricker AD, Stombaugh J, Knight R, Angenent LT, Ley RE. Succession of microbial consortia in the developing infant gut microbiome. Proc Natl Acad Sci U S A. 2011 Mar 15;108 Suppl 1(Suppl 1):4578-85. doi: 10.1073/pnas.1000081107. Epub 2010 Jul 28. PMID 20668239
- [Background] Kostic AD, Chun E, Robertson L, Glickman JN, Gallini CA, Michaud M, Clancy TE, Chung DC, Lochhead P, Hold GL, El-Omar EM, Brenner D, Fuchs CS, Meyerson M, Garrett WS. Fusobacterium nucleatum potentiates intestinal tumorigenesis and modulates the tumor-immune microenvironment. Cell Host Microbe. 2013 Aug 14;14(2):207-15. doi: 10.1016/j.chom.2013.07.007. PMID 23954159
- [Background] Locey KJ, Lennon JT. Scaling laws predict global microbial diversity. Proc Natl Acad Sci U S A. 2016 May 24;113(21):5970-5. doi: 10.1073/pnas.1521291113. Epub 2016 May 2. PMID 27140646
- [Background] Lozupone CA, Stombaugh JI, Gordon JI, Jansson JK, Knight R. Diversity, stability and resilience of the human gut microbiota. Nature. 2012 Sep 13;489(7415):220-30. doi: 10.1038/nature11550. PMID 22972295
- [Background] Lu J, Hu S, Miccoli P, Zeng Q, Liu S, Ran L, Hu C. Non-invasive diagnosis of papillary thyroid microcarcinoma: a NMR-based metabolomics approach. Oncotarget. 2016 Dec 6;7(49):81768-81777. doi: 10.18632/oncotarget.13178. PMID 27835583
- [Background] Maier TV, Lucio M, Lee LH, VerBerkmoes NC, Brislawn CJ, Bernhardt J, Lamendella R, McDermott JE, Bergeron N, Heinzmann SS, Morton JT, Gonzalez A, Ackermann G, Knight R, Riedel K, Krauss RM, Schmitt-Kopplin P, Jansson JK. Impact of Dietary Resistant Starch on the Human Gut Microbiome, Metaproteome, and Metabolome. mBio. 2017 Oct 17;8(5):e01343-17. doi: 10.1128/mBio.01343-17. PMID 29042495
- [Background] Masetti G, Moshkelgosha S, Kohling HL, Covelli D, Banga JP, Berchner-Pfannschmidt U, Horstmann M, Diaz-Cano S, Goertz GE, Plummer S, Eckstein A, Ludgate M, Biscarini F, Marchesi JR; INDIGO consortium. Gut microbiota in experimental murine model of Graves' orbitopathy established in different environments may modulate clinical presentation of disease. Microbiome. 2018 May 25;6(1):97. doi: 10.1186/s40168-018-0478-4. PMID 29801507
- [Background] Ni J, Shen TD, Chen EZ, Bittinger K, Bailey A, Roggiani M, Sirota-Madi A, Friedman ES, Chau L, Lin A, Nissim I, Scott J, Lauder A, Hoffmann C, Rivas G, Albenberg L, Baldassano RN, Braun J, Xavier RJ, Clish CB, Yudkoff M, Li H, Goulian M, Bushman FD, Lewis JD, Wu GD. A role for bacterial urease in gut dysbiosis and Crohn's disease. Sci Transl Med. 2017 Nov 15;9(416):eaah6888. doi: 10.1126/scitranslmed.aah6888. PMID 29141885
- [Background] Nikiforov YE, Steward DL, Robinson-Smith TM, Haugen BR, Klopper JP, Zhu Z, Fagin JA, Falciglia M, Weber K, Nikiforova MN. Molecular testing for mutations in improving the fine-needle aspiration diagnosis of thyroid nodules. J Clin Endocrinol Metab. 2009 Jun;94(6):2092-8. doi: 10.1210/jc.2009-0247. Epub 2009 Mar 24. PMID 19318445
- [Background] O'Toole PW. Changes in the intestinal microbiota from adulthood through to old age. Clin Microbiol Infect. 2012 Jul;18 Suppl 4:44-6. doi: 10.1111/j.1469-0691.2012.03867.x. PMID 22647048
- [Background] Sancho JJ, Lennard TW, Paunovic I, Triponez F, Sitges-Serra A. Prophylactic central neck disection in papillary thyroid cancer: a consensus report of the European Society of Endocrine Surgeons (ESES). Langenbecks Arch Surg. 2014 Feb;399(2):155-63. doi: 10.1007/s00423-013-1152-8. Epub 2013 Dec 19. PMID 24352594
- [Background] Virili C, Fallahi P, Antonelli A, Benvenga S, Centanni M. Gut microbiota and Hashimoto's thyroiditis. Rev Endocr Metab Disord. 2018 Dec;19(4):293-300. doi: 10.1007/s11154-018-9467-y. PMID 30294759
- [Background] Vought RL, Brown FA, Sibinovic KH, McDaniel EG. Effect of changing intestinal bacterial flora on thyroid function in the rat. Horm Metab Res. 1972 Jan;4(1):43-7. doi: 10.1055/s-0028-1094095. No abstract available. PMID 4110893
- [Background] Wada N, Duh QY, Sugino K, Iwasaki H, Kameyama K, Mimura T, Ito K, Takami H, Takanashi Y. Lymph node metastasis from 259 papillary thyroid microcarcinomas: frequency, pattern of occurrence and recurrence, and optimal strategy for neck dissection. Ann Surg. 2003 Mar;237(3):399-407. doi: 10.1097/01.SLA.0000055273.58908.19. PMID 12616125
- [Background] Zhang J, Zhang F, Zhao C, Xu Q, Liang C, Yang Y, Wang H, Shang Y, Wang Y, Mu X, Zhu D, Zhang C, Yang J, Yao M, Zhang L. Dysbiosis of the gut microbiome is associated with thyroid cancer and thyroid nodules and correlated with clinical index of thyroid function. Endocrine. 2019 Jun;64(3):564-574. doi: 10.1007/s12020-018-1831-x. Epub 2018 Dec 24. PMID 30584647
- [Background] Zhao F, Feng J, Li J, Zhao L, Liu Y, Chen H, Jin Y, Zhu B, Wei Y. Alterations of the Gut Microbiota in Hashimoto's Thyroiditis Patients. Thyroid. 2018 Feb;28(2):175-186. doi: 10.1089/thy.2017.0395. Epub 2018 Feb 1. PMID 29320965
- [Background] Zhao Q, Ming J, Liu C, Shi L, Xu X, Nie X, Huang T. Multifocality and total tumor diameter predict central neck lymph node metastases in papillary thyroid microcarcinoma. Ann Surg Oncol. 2013 Mar;20(3):746-52. doi: 10.1245/s10434-012-2654-2. Epub 2012 Sep 13. PMID 22972508
- [Background] Zhou L, Li X, Ahmed A, Wu D, Liu L, Qiu J, Yan Y, Jin M, Xin Y. Gut microbe analysis between hyperthyroid and healthy individuals. Curr Microbiol. 2014 Nov;69(5):675-80. doi: 10.1007/s00284-014-0640-6. Epub 2014 Jun 27. PMID 24969306